CLINICAL TRIAL: NCT07020780
Title: Five Fractions Ultrahypofractionated Whole Breast Radiotherapy and Simultaneous Integrated Boost to the Tumor Bed, for Breast Cancer Patients With Unfavorable Characteristics
Brief Title: 5 fr Ultrahypofractionated WBI and SIB for Breast Cancer With Unfavorable Characteristics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrei Fodor, MD, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HY FIVE
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Whole Breast Irradiation; Simultaneous Integrated Boost; Adjuvant Radiotherapy; Utrahypofractionated Radiotherapy; Moderately Hypofractionated Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 458 patients are expected to be enrolled in this prospective, randomized study. A power of 80% and a significance level α of 5% are used to calculate the sample size. The hypothesis is that the proportion of patients free from local recurrence 5 years after the end of treatment is not less than 95.4%, with a margin of 5%. A total of 218 patients per arm are needed, and an additional 5% (22 patients) to compensate for dropouts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Five fractions radiotherapy (Experimental): Patients in the study (randomized to arm 1) will be treated to the whole breast to a total dose (TD) of 26 Gy in 5 fractions, with simultaneous integrated boost (SIB) to a TD of 30 Gy to the tumor bed. For each patient, an IMRT (intensity modulated radiotherapy) treatment plan will be created to ensure adequate coverage of the treatment volumes and the tolerability of the Organs At Risk (OAR). Specific, already validated dose-volume constraints will be applied for the evaluation of OARs. The dose-volume histogram (DVH) for the Gross Tumor Volume (GTV), Clinical Target Volume (CTV), PTV, and OAR will be calculated in order to achieve the best optimization in terms of tolerability and efficacy.
  Interventions: Radiation: Adjuvant 5 fractions whole breast irradiation with simultaneous integrated boost to the tumor bed
- Arm 2- Fifteen fractions radiotherapy (Active Comparator): Patients randomized to arm 2 will be treated according to the standard protocol of our department, delivering adjuvant whole breast irradiation (WBI) to a total dose (TD) of 40.05 Gy in 15 fractions, with simultaneous integrated boost (SIB) to the tumor bed to a TD of 48 Gy.
  Interventions: Radiation: Adjuvant 5 fractions whole breast irradiation with simultaneous integrated boost to the tumor bed

INTERVENTIONS:
Radiation: Adjuvant 5 fractions whole breast irradiation with simultaneous integrated boost to the tumor bed — Experimental arm (arm 1-five fractions WBI) patients will be treated to a total dose (TD) of 26 Gy in 5 fractions to whole breast, and a simultaneous integrated boost (SIB) to a TD of 30 Gy to the tumor bed, while arm 2-fifteen-fractions WBI patients with 40 Gy/15 fractions to PTV, and 48 Gy SIB to the tumor bed.
  Other Names: Ultrahypofractionated WBI with SIB

SUMMARY:
This is a prospective, randomized, single-center, non-inferiority interventional clinical trial comparing whole breast irradiation (WBI) to a total dose of 26 Gy in 5 fractions with simultaneous integrated boost (SIB) to the tumor bed to a total dose of 30 Gy, and WBI to a total dose of 40.05 Gy in 15 fractions with SIB to the tumor bed to a total dose of 48 Gy (standard treatment), for young or unfavorable breast cancer patients.

DETAILED DESCRIPTION:
The project refers to a study on patients with T1-T3 Nx-N3 breast cancer, aged under 40 years or with unfavorable histology (lobular carcinoma, multifocal tumor, or histological subtypes Luminal B Her2 positive, Hormonal Receptors negative Her 2 positive, Triple Negative Breast Cancer-TNBC-) treated with breast-conserving surgery (BCS) and radiotherapy to the whole breast (+/- lymph node areas) to a total dose of 26 Gy in 5 fractions, with simultaneous boost (SIB) to the tumor bed to the total dose of 30 Gy, that will be compared with the current departmental standard of moderately hypofractionated radiotherapy to the whole breast, to 40.05 Gy in 15 fractions, with SIB to the tumor bed to a total dose of 48 Gy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of breast cancer
2. Patients younger than 40 years regardless of histological subtype, or patients between 40 and 70 years with lobular carcinoma, histological subtypes Luminal B Her2 positive, or with hormone receptors negative and Her2 positive (ErbB2), or triple negative (TNBC)
3. Signed informed consent
4. Clinical stage T1-T3, Nx-N3
5. Negative surgical margins (≥ 0.2 cm)
6. Clinical M0 in the previous 3 months
7. PS (ECOG) ≤2
8. No previous thoracic radiotherapy
9. Fertile women using contraceptive methods started during oncological treatment

Exclusion Criteria:

1. Patients with favorable characteristics (Luminal A, Luminal B Her2 negative, ≥ 40 years) undergoing partial irradiation
2. Patients who have undergone mastectomy
3. Multicentric tumors
4. Positive or close surgical margins (<0.2 cm)
5. BRCA1/2 positive (only if known)
6. Serious systemic diseases
7. Mental or other disorders that may prevent the patient from signing the informed consent
8. Previous invasive tumor, except skin cancer (excluding melanoma) unless the patient has been disease-free for at least 3 years (for example carcinoma in situ of the oral cavity or bladder)
9. Collagen or autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, scleroderma, Sjogren's syndrome)
10. Evidence of distant metastases (M1)
11. Contraindication to treatment systemic
12. Pregnant women
13. Non-compliance with the dose limits established in the treatment plan

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with breast cancer and age <40 years regardless if histology, or 40-70 years old with unfavorable characteristics.
Enrollment: 458 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Local Relapse Free Survival (LRFS) | 5 years
  o demonstrate the non-inferiority of local control (local relapse free survival - LRFS) of the study treatment (delivered in five fractions) compared to the department's standard WBI treatment (delivered in 15 fractions).

SECONDARY OUTCOMES:
Acute toxicity | 1 month
  Acute toxicity grade ≥3 as the maximum toxicity value within 1 month and 3 months after the completion of radiotherapy treatment evaluated with RTOG/EORTC scale with 4 grades, from 0 no change to 4, worst toxicity
Acute toxicity | 3 months
  Acute toxicity grade ≥3 as the maximum toxicity value within 1 month and 3 months after the completion of radiotherapy treatment evaluated with RTOG/EORTC scale with 4 grades, from 0 no change to 4, worst toxicity
Late toxicity | 5 years
  Late skin toxicity evaluated with RTOG/EORTC scale, with 4 grades, from 0 = no change, to 4 = maximum toxicity
Late toxicity | 5 years
  Late toxicity evaluated with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, with 5 grades, from 0 = no change, to 5 = death for toxicity
Local Control | 5 years
  Local control of the treated site expressed in terms of local recurrence rate
Ipsilateral Breast Tumor Recurrence (IBTR) | 5 years
  Ipsilateral breast tumor recurrence - IBTR- of the study treatment (delivered in 5 fractions WBI+SIB) compared to the department's standard WBI+SIB treatment (delivered in 15 fractions).
Regional Relapse-Free Survival (RRFS) | From the date of radiotherapy end until the date of regional relapse, assessed up to 5 years
  Time to regional (nodal) recurrence
Distant Metastasis-Free Survival (DMFS) | From the date of radiotherapy end until the date of distant metasis diagnosis, assessed up to 5 years
  Time to distant (metastatic) relapse
Disease-Free Survival (DFS) | From the date of radiotherapy end until the date of first, any ( local, regional, distant) relapse, assessed up to 5 years
  Time to first any relapse: local, regional or distant
Breast Cancer Specific Survival (BCSS) | From the date of radiotherapy end until the date of death from breast cancer, assessed up to 5 years
  Time until death from breast cancer
Overall Survival (OS) | From the date of radiotherapy end until the date of death from any cause, assessed up to 5 years
  Time until death from any cause
Cosmesis | 5 years
  Cosmetic results evaluated with Harvard scale. It assesses the global esthetic appearance of the breast, categorized as Excellent, Good, Fair, or Poor
Acute toxicity interim analysis | 3 months
  An interim analysis of acute toxicity (with RTOG/EORTC andf CTCAE v5.0 scales) will be performed for the first 200 patients
Late toxicity interim analysis | 42 months
  An interim analysis of late toxicity (with RTOG/EORTC andf CTCAE v5.0 scales) will be performed for the first 200 patients
Local relapse interim analysis | 42 months
  An interim analysis of local relapse rate will be performed for the first 200 patients
Incidence of Treatment-Emergent Adverse Events as assessed with breast tumor specific quality of life questionnaires | 5 years
  Survey with the questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) Quality of life of brain tumor patients (EORTC QLQ BR42) which contains 42 questions on patients' quality of life with answers from 1, lowest grade, to 4, highest grade
Modeling of organ movement | 15 days
  Modeling of organ movement during treatment
Radiomics | 5 years
  CT radiomic features predicting relapse or death will be extracted, acording to IBSI (Image Biomarker Standardisation Initiative), owning to the different families of features: Morphology, Statistical, Intensity Histogram, Grey Level Cooccurrence Matrix 3D-average, Grey Level Co-occurrence Matrix 3D-combined, Grey Level Run Lenght 3D-average. Grey Level Run Lenght 3D_combined, Grey Level Size Zone Matrix 3D, Neighbors Grey Tone Difference Matrix 3D, Grey Level Distance Zone Matrix 3D, standard convolutional filters within radiomic workflow (wavelets, Laplacian of Gaussian). Area Under Curve (AUC) will be taken as representative of the discriminative power for each of the significant RF.
Predictive factors for toxicity | 5 years
  Identification of clinical, imaging, and laboratory prognostic factors for toxicity. Univariable and multivariable Cox analysis will be performed to identify factors associated with >/= G2 toxicity
Predictive factors for disease progression | 5 years
  Identification of clinical, imaging, and laboratory prognostic factors for an aggressive phenotype of breast cancer. Univariable and multivariable analysis will be performed to identify factors associated with disease progression
Predictive factors for death | 5 years
  Identification of clinical, imaging, and laboratory prognostic factors for an aggressive phenotype of breast cancer. Univariable and multivariable Cox analysis will be performed to identify factors associated with death.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Fodor, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author will be evaluated by the Lombardy Territorial Ethics Committee 1
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for 5 years after the end of the study
Access Criteria: request from the corresponding author approved by the Lombardy Territorial Ethics Committee

REFERENCES:
- [Result] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Result] Clark RM, Whelan T, Levine M, Roberts R, Willan A, McCulloch P, Lipa M, Wilkinson RH, Mahoney LJ. Randomized clinical trial of breast irradiation following lumpectomy and axillary dissection for node-negative breast cancer: an update. Ontario Clinical Oncology Group. J Natl Cancer Inst. 1996 Nov 20;88(22):1659-64. doi: 10.1093/jnci/88.22.1659. PMID 8931610
- [Result] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Result] Shaitelman SF, Lei X, Thompson A, Schlembach P, Bloom ES, Arzu IY, Buchholz D, Chronowski G, Dvorak T, Grade E, Hoffman K, Perkins G, Reed VK, Shah SJ, Stauder MC, Strom EA, Tereffe W, Woodward WA, Amaya DN, Shen Y, Hortobagyi GN, Hunt KK, Buchholz TA, Smith BD. Three-Year Outcomes With Hypofractionated Versus Conventionally Fractionated Whole-Breast Irradiation: Results of a Randomized, Noninferiority Clinical Trial. J Clin Oncol. 2018 Oct 31;36(35):JCO1800317. doi: 10.1200/JCO.18.00317. Online ahead of print. PMID 30379626
- [Result] Chua BH, Link EK, Kunkler IH, Whelan TJ, Westenberg AH, Gruber G, Bryant G, Ahern V, Purohit K, Graham PH, Akra M, McArdle O, O'Brien P, Harvey JA, Kirkove C, Maduro JH, Campbell ID, Delaney GP, Martin JD, Vu TTT, Muanza TM, Neal A, Olivotto IA; BIG 3-07/TROG 07.01 trial investigators. Radiation doses and fractionation schedules in non-low-risk ductal carcinoma in situ in the breast (BIG 3-07/TROG 07.01): a randomised, factorial, multicentre, open-label, phase 3 study. Lancet. 2022 Aug 6;400(10350):431-440. doi: 10.1016/S0140-6736(22)01246-6. PMID 35934006
- [Result] Meattini I, Becherini C, Boersma L, Kaidar-Person O, Marta GN, Montero A, Offersen BV, Aznar MC, Belka C, Brunt AM, Dicuonzo S, Franco P, Krause M, MacKenzie M, Marinko T, Marrazzo L, Ratosa I, Scholten A, Senkus E, Stobart H, Poortmans P, Coles CE. European Society for Radiotherapy and Oncology Advisory Committee in Radiation Oncology Practice consensus recommendations on patient selection and dose and fractionation for external beam radiotherapy in early breast cancer. Lancet Oncol. 2022 Jan;23(1):e21-e31. doi: 10.1016/S1470-2045(21)00539-8. PMID 34973228
- [Result] Marta GN, Coles C, Kaidar-Person O, Meattini I, Hijal T, Zissiadis Y, Pignol JP, Ramiah D, Ho AY, Cheng SH, Sancho G, Offersen BV, Poortmans P. The use of moderately hypofractionated post-operative radiation therapy for breast cancer in clinical practice: A critical review. Crit Rev Oncol Hematol. 2020 Dec;156:103090. doi: 10.1016/j.critrevonc.2020.103090. Epub 2020 Aug 26. PMID 33091800
- [Result] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Result] Coles CE, Haviland JS, Kirby AM, Griffin CL, Sydenham MA, Titley JC, Bhattacharya I, Brunt AM, Chan HYC, Donovan EM, Eaton DJ, Emson M, Hopwood P, Jefford ML, Lightowlers SV, Sawyer EJ, Syndikus I, Tsang YM, Twyman NI, Yarnold JR, Bliss JM; IMPORT Trial Management Group. Dose-escalated simultaneous integrated boost radiotherapy in early breast cancer (IMPORT HIGH): a multicentre, phase 3, non-inferiority, open-label, randomised controlled trial. Lancet. 2023 Jun 24;401(10394):2124-2137. doi: 10.1016/S0140-6736(23)00619-0. Epub 2023 Jun 8. PMID 37302395
- [Result] Haviland JS, Bentzen SM, Bliss JM, Yarnold JR; START Trial Management Group. Prolongation of overall treatment time as a cause of treatment failure in early breast cancer: An analysis of the UK START (Standardisation of Breast Radiotherapy) trials of radiotherapy fractionation. Radiother Oncol. 2016 Dec;121(3):420-423. doi: 10.1016/j.radonc.2016.08.027. Epub 2016 Sep 22. PMID 27666929
- [Result] Lievens Y. Hypofractionated breast radiotherapy: financial and economic consequences. Breast. 2010 Jun;19(3):192-7. doi: 10.1016/j.breast.2010.03.003. PMID 20511069
- [Result] Marta GN, Ramiah D, Kaidar-Person O, Kirby A, Coles C, Jagsi R, Hijal T, Sancho G, Zissiadis Y, Pignol JP, Ho AY, Cheng SH, Offersen BV, Meattini I, Poortmans P. The Financial Impact on Reimbursement of Moderately Hypofractionated Postoperative Radiation Therapy for Breast Cancer: An International Consortium Report. Clin Oncol (R Coll Radiol). 2021 May;33(5):322-330. doi: 10.1016/j.clon.2020.12.008. Epub 2020 Dec 23. PMID 33358283
- [Result] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Result] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Result] Lewis P, Brunt AM, Coles C, Griffin S, Locke I, Roques T; Breast Radiotherapy Consensus Working Group. Moving Forward Fast with FAST-Forward. Clin Oncol (R Coll Radiol). 2021 Jul;33(7):427-429. doi: 10.1016/j.clon.2021.04.007. Epub 2021 May 14. No abstract available. PMID 33994270
- [Result] Montero A, Ciervide R, Canadillas C, Alvarez B, Garcia-Aranda M, Alonso R, Lopez M, Chen-Zhao X, Alonso L, Valero J, Sanchez E, Hernando O, Garcia de Acilu P, Fernandez-Leton P, Rubio C. Acute skin toxicity of ultra-hypofractionated whole breast radiotherapy with simultaneous integrated boost for early breast cancer. Clin Transl Radiat Oncol. 2023 Jun 15;41:100651. doi: 10.1016/j.ctro.2023.100651. eCollection 2023 Jul. PMID 37388711
- [Result] Monten C, Lievens Y, Olteanu LAM, Paelinck L, Speleers B, Deseyne P, Van Den Broecke R, De Neve W, Veldeman L. Highly Accelerated Irradiation in 5 Fractions (HAI-5): Feasibility in Elderly Women With Early or Locally Advanced Breast Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):922-930. doi: 10.1016/j.ijrobp.2017.01.229. Epub 2017 Feb 1. PMID 28366576
- [Result] Van Hulle H, Vakaet V, Monten C, Deseyne P, Schoepen M, Colman C, Paelinck L, Van Greveling A, Post G, Speleers B, Vandecasteele K, Mareel M, De Neve W, Veldeman L. Acute toxicity and health-related quality of life after accelerated whole breast irradiation in 5 fractions with simultaneous integrated boost. Breast. 2021 Feb;55:105-111. doi: 10.1016/j.breast.2020.12.009. Epub 2020 Dec 24. PMID 33401157
- [Result] Boccardi M, Cilla S, Fanelli M, Romano C, Bonome P, Ferro M, Pezzulla D, Di Marco R, Deodato F, Macchia G. Ultra-Hypofractionated Whole Breast Radiotherapy with Automated Hybrid-VMAT Technique: A Pilot Study on Safety, Skin Toxicity and Aesthetic Outcomes. Breast Cancer (Dove Med Press). 2024 Sep 16;16:611-619. doi: 10.2147/BCTT.S470417. eCollection 2024. PMID 39310783
- [Result] Coles CE, Aristei C, Bliss J, Boersma L, Brunt AM, Chatterjee S, Hanna G, Jagsi R, Kaidar Person O, Kirby A, Mjaaland I, Meattini I, Luis AM, Marta GN, Offersen B, Poortmans P, Rivera S. International Guidelines on Radiation Therapy for Breast Cancer During the COVID-19 Pandemic. Clin Oncol (R Coll Radiol). 2020 May;32(5):279-281. doi: 10.1016/j.clon.2020.03.006. No abstract available. PMID 32241520
- [Result] Meattini I, Palumbo I, Becherini C, Borghesi S, Cucciarelli F, Dicuonzo S, Fiorentino A, Spoto R, Poortmans P, Aristei C, Livi L. The Italian Association for Radiotherapy and Clinical Oncology (AIRO) position statements for postoperative breast cancer radiation therapy volume, dose, and fractionation. Radiol Med. 2022 Dec;127(12):1407-1411. doi: 10.1007/s11547-022-01563-9. Epub 2022 Oct 6. PMID 36201098
- [Result] Brunt AM, Haviland JS, Wheatley DA, Sydenham MA, Bloomfield DJ, Chan C, Cleator S, Coles CE, Donovan E, Fleming H, Glynn D, Goodman A, Griffin S, Hopwood P, Kirby AM, Kirwan CC, Nabi Z, Patel J, Sawyer E, Somaiah N, Syndikus I, Venables K, Yarnold JR, Bliss JM; FAST-Forward Trial Management Group. One versus three weeks hypofractionated whole breast radiotherapy for early breast cancer treatment: the FAST-Forward phase III RCT. Health Technol Assess. 2023 Nov;27(25):1-176. doi: 10.3310/WWBF1044. PMID 37991196
- [Result] Chatterjee S, Chakraborty S; HYPORT Adjuvant Author Group. Hypofractionated radiation therapy comparing a standard radiotherapy schedule (over 3 weeks) with a novel 1-week schedule in adjuvant breast cancer: an open-label randomized controlled study (HYPORT-Adjuvant)-study protocol for a multicentre, randomized phase III trial. Trials. 2020 Sep 30;21(1):819. doi: 10.1186/s13063-020-04751-y. PMID 32998747
- [Result] Chakraborty S, Chatterjee S; Hyport Adjuvant Author Group. HYPORT adjuvant acute toxicity and patient dosimetry quality assurance results - Interim analysis. Radiother Oncol. 2022 Sep;174:59-68. doi: 10.1016/j.radonc.2022.07.003. Epub 2022 Jul 9. PMID 35817323
- [Result] Ratosa I, Montero A, Ciervide R, Alvarez B, Garcia-Aranda M, Valero J, Chen-Zhao X, Lopez M, Zucca D, Hernando O, Sanchez E, de la Casa MA, Alonso R, Fernandez-Leton P, Rubio C. Ultra-hypofractionated one-week locoregional radiotherapy for patients with early breast cancer: Acute toxicity results. Clin Transl Radiat Oncol. 2024 Mar 13;46:100764. doi: 10.1016/j.ctro.2024.100764. eCollection 2024 May. PMID 38516338
- [Result] Yadav BS, Dey T. Hypofractionation for Regional Nodal Irradiation in Breast Cancer: Best of Both the Worlds. Clin Breast Cancer. 2024 Jul;24(5):399-410. doi: 10.1016/j.clbc.2024.03.007. Epub 2024 Mar 14. PMID 38614852
- [Result] Boyages J, Harris JR. Local therapy of invasive disease. Hematol Oncol Clin North Am. 1989 Dec;3(4):675-90. PMID 2691494
- [Result] Mannino M, Yarnold J. Accelerated partial breast irradiation trials: diversity in rationale and design. Radiother Oncol. 2009 Apr;91(1):16-22. doi: 10.1016/j.radonc.2008.12.011. Epub 2009 Jan 27. PMID 19178972
- [Result] Holland R, Connolly JL, Gelman R, Mravunac M, Hendriks JH, Verbeek AL, Schnitt SJ, Silver B, Boyages J, Harris JR. The presence of an extensive intraductal component following a limited excision correlates with prominent residual disease in the remainder of the breast. J Clin Oncol. 1990 Jan;8(1):113-8. doi: 10.1200/JCO.1990.8.1.113. PMID 2153190
- [Result] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Result] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Result] Bartelink H, Maingon P, Poortmans P, Weltens C, Fourquet A, Jager J, Schinagl D, Oei B, Rodenhuis C, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan D, Dubois JB, Remouchamps V, Mirimanoff RO, Collette S, Collette L; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):47-56. doi: 10.1016/S1470-2045(14)71156-8. Epub 2014 Dec 9. PMID 25500422
- [Result] Fodor A, Brombin C, Mangili P, Borroni F, Pasetti M, Tummineri R, Zerbetto F, Longobardi B, Perna L, Dell'Oca I, Deantoni CL, Deli AM, Chiara A, Broggi S, Castriconi R, Esposito PG, Slim N, Passoni P, Baroni S, Villa SL, Rancoita PMV, Fiorino C, Del Vecchio A, Bianchini G, Gentilini OD, Di Serio MS, Di Muzio NG. Impact of molecular subtype on 1325 early-stage breast cancer patients homogeneously treated with hypofractionated radiotherapy without boost: Should the indications for radiotherapy be more personalized? Breast. 2021 Feb;55:45-54. doi: 10.1016/j.breast.2020.12.004. Epub 2020 Dec 9. PMID 33326894
- [Result] Whelan TJ, Kim DH, Sussman J. Clinical experience using hypofractionated radiation schedules in breast cancer. Semin Radiat Oncol. 2008 Oct;18(4):257-64. doi: 10.1016/j.semradonc.2008.04.008. PMID 18725113
- [Result] Qi XS, White J, Li XA. Is alpha/beta for breast cancer really low? Radiother Oncol. 2011 Aug;100(2):282-8. doi: 10.1016/j.radonc.2011.01.010. Epub 2011 Feb 28. PMID 21367477
- [Result] Ray KJ, Sibson NR, Kiltie AE. Treatment of Breast and Prostate Cancer by Hypofractionated Radiotherapy: Potential Risks and Benefits. Clin Oncol (R Coll Radiol). 2015 Jul;27(7):420-6. doi: 10.1016/j.clon.2015.02.008. Epub 2015 Mar 7. PMID 25752244
- [Result] Brand DH, Kirby AM, Yarnold JR, Somaiah N. How Low Can You Go? The Radiobiology of Hypofractionation. Clin Oncol (R Coll Radiol). 2022 May;34(5):280-287. doi: 10.1016/j.clon.2022.02.009. Epub 2022 Mar 5. PMID 35260319
- [Result] van Leeuwen CM, Oei AL, Crezee J, Bel A, Franken NAP, Stalpers LJA, Kok HP. The alfa and beta of tumours: a review of parameters of the linear-quadratic model, derived from clinical radiotherapy studies. Radiat Oncol. 2018 May 16;13(1):96. doi: 10.1186/s13014-018-1040-z. PMID 29769103
- [Result] Schneider U, Besserer J, Mack A. Hypofractionated radiotherapy has the potential for second cancer reduction. Theor Biol Med Model. 2010 Feb 11;7:4. doi: 10.1186/1742-4682-7-4. PMID 20149259
- [Result] Dasu A, Toma-Dasu I, Olofsson J, Karlsson M. The use of risk estimation models for the induction of secondary cancers following radiotherapy. Acta Oncol. 2005;44(4):339-47. doi: 10.1080/02841860510029833. PMID 16120542
- [Result] Berrington de Gonzalez A, Gilbert E, Curtis R, Inskip P, Kleinerman R, Morton L, Rajaraman P, Little MP. Second solid cancers after radiation therapy: a systematic review of the epidemiologic studies of the radiation dose-response relationship. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):224-33. doi: 10.1016/j.ijrobp.2012.09.001. Epub 2012 Oct 24. PMID 23102695
- [Result] Sitathanee C, Tangboonduangjit P, Dhanachai M, Suntiwong S, Yongvithisatid P, Rutchantuk S, Changkaew P, Watjiranon R, Khachonkham S, Boonkitticharoen V. Secondary cancer risk from modern external-beam radiotherapy of prostate cancer patients: Impact of fractionation and dose distribution. J Radiat Res. 2021 Jul 10;62(4):707-717. doi: 10.1093/jrr/rrab038. PMID 33993271
- [Result] Ciabattoni A, Gregucci F, De Rose F, Falivene S, Fozza A, Daidone A, Morra A, Smaniotto D, Barbara R, Lozza L, Vidali C, Borghesi S, Palumbo I, Huscher A, Perrucci E, Baldissera A, Tolento G, Rovea P, Franco P, De Santis MC, Grazia AD, Marino L, Meduri B, Cucciarelli F, Aristei C, Bertoni F, Guenzi M, Leonardi MC, Livi L, Nardone L, De Felice F, Rosetto ME, Mazzuoli L, Anselmo P, Arcidiacono F, Barbarino R, Martinetti M, Pasinetti N, Desideri I, Marazzi F, Ivaldi G, Bonzano E, Cavallari M, Cerreta V, Fusco V, Sarno L, Bonanni A, Mangiacotti MG, Prisco A, Buonfrate G, Andrulli D, Fontana A, Bagnoli R, Marinelli L, Reverberi C, Scalabrino G, Corazzi F, Doino D, Di Genesio-Pagliuca M, Lazzari M, Mascioni F, Pace MP, Mazza M, Vitucci P, Spera A, Macchia G, Boccardi M, Evangelista G, Sola B, La Porta MR, Fiorentino A, Levra NG, Ippolito E, Silipigni S, Osti MF, Mignogna M, Alessandro M, Ursini LA, Nuzzo M, Meattini I, D'Ermo G. AIRO Breast Cancer Group Best Clinical Practice 2022 Update. Tumori. 2022 Jul;108(2_suppl):1-144. doi: 10.1177/03008916221088885. PMID 36112842
- [Result] Offersen BV, Boersma LJ, Kirkove C, Hol S, Aznar MC, Biete Sola A, Kirova YM, Pignol JP, Remouchamps V, Verhoeven K, Weltens C, Arenas M, Gabrys D, Kopek N, Krause M, Lundstedt D, Marinko T, Montero A, Yarnold J, Poortmans P. ESTRO consensus guideline on target volume delineation for elective radiation therapy of early stage breast cancer. Radiother Oncol. 2015 Jan;114(1):3-10. doi: 10.1016/j.radonc.2014.11.030. Epub 2015 Jan 24. PMID 25630428
- [Result] Duane F, Aznar MC, Bartlett F, Cutter DJ, Darby SC, Jagsi R, Lorenzen EL, McArdle O, McGale P, Myerson S, Rahimi K, Vivekanandan S, Warren S, Taylor CW. A cardiac contouring atlas for radiotherapy. Radiother Oncol. 2017 Mar;122(3):416-422. doi: 10.1016/j.radonc.2017.01.008. Epub 2017 Feb 21. PMID 28233564